CLINICAL TRIAL: NCT06284148
Title: EHR-based Screening and Intervention for Intimate Partner Violence
Brief Title: Confidential IPV Screening Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Leslie Lenert, Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: Pro00093964; 5R18HS025654-03 (AHRQ)
Record Dates: First submitted 2024-02-09; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Violence, Domestic
Keywords: Intimate Partner Violence
MeSH Terms: interventions — Mass Screening; Restraint, Physical; Referral and Consultation

STUDY DESIGN:
Intervention Model Description: This is a stepped wedge cluster randomized trial which has 3 sequences starting intervention in randomized order.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sequence 1 (Other): 5 clinics. In stepped wedge design study, this was the sequence with shortest control (run-in) period.
  All sequences have a run-in period and intervention period. In control period participants were screened using existing nurse-led oral screening, in intervention period both - nurse-led and our new confidential screen were used at the same time.
  Interventions: Diagnostic Test: Screening for intimate partner violence; Other: Assessment and referral
- Sequence 2 (Other): 5 clinics.
  Interventions: Diagnostic Test: Screening for intimate partner violence; Other: Assessment and referral
- Sequence 3 (Other): 5 clinics. This was the sequence with longest control (run-in) period.
  Interventions: Diagnostic Test: Screening for intimate partner violence; Other: Assessment and referral

INTERVENTIONS:
Diagnostic Test: Screening for intimate partner violence — confidential screening using exam computer
Other: Assessment and referral — confidential assessment and referral of high-risk patients using decision-support templates

SUMMARY:
Intimate partner violence (IPV) against women in the US is a serious public health problem and a human rights issue. Our research team has developed confidential screening tools using exam-room computer for intimate partner violence to be used in primary care.

DETAILED DESCRIPTION:
The objective of this study was to develop and evaluate an integrated suite of electronic health record (EHR) tools that automates "best practices" from Northern California Kaiser Permanente for screening and intervention for IPV identified within clinical settings. The goal of the intervention goes beyond mere screening of patients for IPV and includes tools for assessment of IPV risk, for documentation of IPV care, and support for a warm hand-off during the primary care visit to a national IPV hotline resource. Importantly, the study includes work to keep notes documenting IPV and billing for IPV care confidential, segmenting this care in a secure segment of the electronic health record.

ELIGIBILITY:
Inclusion Criteria:

* Being an Medical University of South Carolina patient at primary care clinics (family medicine)
* Women 18-49 years of age inclusive
* Reported yes to wanting to be contacted for a follow-up research study
* English-speaking

Exclusion Criteria:

* No exclusion criteria

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All patients who identified as women were eligible
Enrollment: 19655 (Actual)
Dates: Start 2010-10-06 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
IPV positive (Yes/No) | 29 months
  Depending on patient's answers to screening questions, they are flagged as either IPV positive or negative
Screening completed (Yes/No) | 29 months
  Whether the assigned screening was completed during patient visit

SECONDARY OUTCOMES:
Severity of risk | 29 months
  using Danger 5 risk assessment, ranging from 0 to 5
Physician compliance with IPV management tools | 29 months
  Measured as the rate of completion of follow-up decision templates, and the rate of referrals for post-visit counseling to a national hotline (a share from screened positive patients

CONTACTS AND LOCATIONS:
Locations (1):
- Biomedical Informatics Center, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Lenert L, Rheingold AA, Simpson KN, Scherbakov D, Aiken M, Hahn C, McCauley JL, Ennis N, Diaz VA. Electronic Health Record-Based Screening for Intimate Partner Violence: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2024 Aug 1;7(8):e2425070. doi: 10.1001/jamanetworkopen.2024.25070. PMID 39088215

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT06284148/Prot_SAP_000.pdf